CLINICAL TRIAL: NCT04133155
Title: Multicenter Retrospective Analysis for Efficacy and Safety of Second-Line Nab-Paclitaxel Plus Gemcitabine After Progression on 1st-line FOLFIRINOX in Advanced Pancreatic Ductal Adenocarcinoma
Brief Title: Retrospective Analysis of 2nd-line Nab-Paclitaxel + Gemcitabine After 1st-line FOLFIRINOX in Pancreatic Cancer
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Collaborators: Bundang CHA Hospital (Other); Ulsan University Hospital (Other)
Responsible Party: Principal Investigator, Changhoon Yoo, Assistant professor, Asan Medical Center
Other Study IDs: AX-NI-PANC-PI-13883
Record Dates: First submitted 2019-10-17; First posted 2019-10-21 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Pancreatic Cancer; Metastatic Pancreatic Cancer
Keywords: Pancreatic cancer; FOLFIRINOX; nab-paclitaxel plus gemcitabine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Taxes; Gemcitabine; Albumin-Bound Paclitaxel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- nab-P + GEM: Nab-paclitaxel plus gemcitabine
  Interventions: Drug: nab paclitaxel plus gemcitabine

INTERVENTIONS:
Drug: nab paclitaxel plus gemcitabine — Nab-paclitaxel 125 mg/m2 weekly for 3 weeks, every 4 weeks Gemcitabine 1000 mg/m2 weekly for 3 weeks, every 4 weeks
  Other Names: Abraxane

SUMMARY:
In this study, clinical data of patients who received 2nd-line Nab-paclitaxel plus Gemcitabine (nab-P+GEM) after progression on 1st-line FOLFIRINOX will be reviewed retrospectively.

DETAILED DESCRIPTION:
FOLFIRINOX is one of standard 1 st-line regimens for patients with advanced PDAC. However, there is no globally established 2 nd-line regimen after the failure of FOLFIRINOX. Although gemcitabine-based regimens are recommended by multiple guidelines and widely used in daily practice, further analysis is needed to reveal the magnitude of clinical benefit with these regimens. Nab-paclitaxel plus Gemcitabine (Nab-P+Gem) is another standard 1 st-line regimen for PDAC, but there are limited data as 2 nd-line therapy in PDAC. Therefore, the investigators are conducting a multicenter retrospective analysis of 2 nd-line nab-P+Gem after progression on FOLFIRINOX in patients with advanced PDAC.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed pancreatic ductal adenocarcinoma
* Administration of 2nd-line nab-paclitaxel plus gemcitabine
* Progression on 1st-line FOLFIRINOX

Exclusion Criteria:

* Pathologic diagnosis other than pancreatic ductal adenocarcinoma
* Administration of nab-paclitaxel plus gemcitabine as 3rd or greater lines of therapy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pathologically confirmed pancreatic ductal adenocarcinoma who received 2nd-line nab-paclitaxel plus gemcitabine after progression on 1st-line FOLFIRINOX
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 1 year
  Time from the start of 2nd-line nab-P + GEM to disease progression or death from any cause, whichever came first

SECONDARY OUTCOMES:
Overall survival | 1 year
  Time from the start of 2nd-line nab-P+GEM to death from any cause
Objective response rates | 1 year
  Tumor response graded by Response Evaluation Criteria in Solid Tumor (RECIST) version 1.1
Toxicity profile | 1 year
  Safety profile graded by National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Changhoon Yoo, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] da Rocha Lino A, Abrahao CM, Brandao RM, Gomes JR, Ferrian AM, Machado MC, Buzaid AC, Maluf FC, Peixoto RD. Role of gemcitabine as second-line therapy after progression on FOLFIRINOX in advanced pancreatic cancer: a retrospective analysis. J Gastrointest Oncol. 2015 Oct;6(5):511-5. doi: 10.3978/j.issn.2078-6891.2015.041. PMID 26487945
- [Background] Kang J, Yoo C, Hwang HS, Hong SM, Kim KP, Kim SY, Hong YS, Kim TW, Ryoo BY. Efficacy and safety of lanreotide in Korean patients with metastatic, well-differentiated gastroenteropancreatic-neuroendocrine tumors: a retrospective analysis. Invest New Drugs. 2019 Aug;37(4):763-770. doi: 10.1007/s10637-018-0710-x. Epub 2018 Dec 10. PMID 30536151
- [Background] Portal A, Pernot S, Siauve N, Landi B, Lepere C, Colussi O, Rougier P, Zaanan A, Verriere B, Taieb J. Sustained response with gemcitabine plus Nab-paclitaxel after folfirinox failure in metastatic pancreatic cancer: report of an effective new strategy. Clin Res Hepatol Gastroenterol. 2014 Apr;38(2):e23-6. doi: 10.1016/j.clinre.2014.01.005. Epub 2014 Feb 18. PMID 24559766
- [Background] Sarabi M, Mais L, Oussaid N, Desseigne F, Guibert P, De La Fouchardiere C. Use of gemcitabine as a second-line treatment following chemotherapy with folfirinox for metastatic pancreatic adenocarcinoma. Oncol Lett. 2017 Jun;13(6):4917-4924. doi: 10.3892/ol.2017.6061. Epub 2017 Apr 20. PMID 28599496
- [Derived] Chae H, Jeong H, Cheon J, Chon HJ, Ryu H, Kim IH, Kang MJ, Jeong JH, Ryoo BY, Kim KP, Yoo C. Efficacy and safety of second-line nab-paclitaxel plus gemcitabine after progression on FOLFIRINOX for unresectable or metastatic pancreatic ductal adenocarcinoma: multicenter retrospective analysis. Ther Adv Med Oncol. 2020 May 27;12:1758835920923424. doi: 10.1177/1758835920923424. eCollection 2020. PMID 32523632